CLINICAL TRIAL: NCT07009171
Title: A Randomized, Double-blind, Placebo-controlled, Dose Finding, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of KDS2010 in Overweight or Obese Patients
Brief Title: Study to Evaluate the Efficacy and Safety of KDS2010 in Overweight or Obese Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBiogen Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB_KDS_OBP2_23; KCT0010560 (Registry Identifier: CRIS)
Record Dates: First submitted 2025-05-15; First posted 2025-06-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Overweight; Obesity; Obese Patients
Keywords: Obese Patients; Overweight; KDS2010; Obesity; MAO-B inhibitor
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Dose-Finding, Phase 2a Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind design is used to ensure scientific validity. Subjects and investigators are unaware of treatment allocation, with identical appearance between the drug and placebo. Randomization numbers are used for subject identification, and group assignments are disclosed only after the end of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1 stage Control Group_Placebo (Placebo Comparator): Administer orally three tablets once daily for 12 weeks (three tablets of 60mg placebo). This group will match the investigational drug in appearance but contain no active ingredients to maintain blinding.
  Interventions: Drug: Placebo
- 1 stage Treatment Group 1_KDS2010 120mg (Experimental): Administer orally three tablets once daily for 12 weeks (two tablets of KDS2010 60mg and one tablet of 60mg placebo). This group will receive the active investigational drug to evaluate its safety and efficacy.
  Interventions: Drug: KDS2010
- 2 stage Control Group_Placebo (Placebo Comparator): Administer orally three tablets once daily for 12 weeks (three tablets of 60mg placebo). This group will match the investigational drug in appearance but contain no active ingredients to maintain blinding.
  Interventions: Drug: Placebo
- 2 stage Treatment Group 1_KDS2010 120mg (Experimental): Administer orally three tablets once daily for 12 weeks (two tablets of KDS2010 60mg and one tablet of 60mg placebo). This group will receive the active investigational drug to evaluate its safety and efficacy.
  Interventions: Drug: KDS2010
- 2 stage Treatment Group 2_KDS2010 180mg (Experimental): Administer orally three tablets once daily for 12 weeks (three tablets of KDS2010 60mg). This group will receive the higher dose of the investigational drug to evaluate its safety and efficacy.
  Interventions: Drug: KDS2010

INTERVENTIONS:
Drug: KDS2010 — KDS2010 will be administered orally once daily, three tablets per day, for 12 weeks. Dosage will be either 120 mg or 180 mg depending on the assigned group.
  Arms: 1 stage Treatment Group 1_KDS2010 120mg; 2 stage Treatment Group 1_KDS2010 120mg; 2 stage Treatment Group 2_KDS2010 180mg
Drug: Placebo — Placebo matching the investigational product in appearance but containing no active ingredient, administered orally once daily, three tablets per day, for 12 weeks.
  Arms: 1 stage Control Group_Placebo; 2 stage Control Group_Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation, Phase 2a study designed to evaluate the safety and efficacy of KDS2010 in overweight or obese patients. Based on preliminary efficacy observed in the Phase 1 study, a multinational clinical trial is being conducted in both Korea and the United States. After a minimum 2-week run-in period, subjects who meet the inclusion and exclusion criteria will be randomized into each dose group at a 2:1 ratio in Stage 1 and in a 1:1:1 ratio in Stage 2, considering stratification by region (Korea/USA).

Subjects will receive the investigational drug for 12 weeks following randomization. Approximately 75 subjects will be enrolled, with 6 subjects in the treatment group and 3 subjects in the control group in Stage 1, and 22 subjects per group in Stage 2.

The primary objectives are to assess the efficacy and safety of KDS2010 in overweight or obese patients. Exploratory objectives include evaluating the proportion of subjects achieving a weight reduction of more than 25% from baseline at Week 12 and assessing changes in MAO-B specific activity and adiponectin levels.

Based on nonclinical and Phase 1 clinical data, KDS2010 will be administered orally once daily at doses of 120 mg and 180 mg throughout the study.

DETAILED DESCRIPTION:
This Phase 2a, multinational, randomized, double-blind, placebo-controlled, dose-finding clinical trial is designed to evaluate the efficacy, safety, and pharmacokinetics of KDS2010, a novel, reversible monoamine oxidase-B (MAO-B) inhibitor, in overweight or obese adult patients. The clinical trial is conducted at selected sites in Korea and the United States.

The study consists of two stages and will enroll approximately 75 subjects. In Stage 1, 9 subjects will be randomized in a 2:1 ratio (KDS2010 120 mg: placebo) to evaluate initial safety and tolerability. Upon completion of the week 13 visit for the last subject in Stage 1, a Safety Review Committee (SRC) will assess cumulative safety data to determine the appropriateness of dose escalation and progression to Stage 2.

If cleared by the SRC, Stage 2 will proceed with 66 subjects randomized equally across three arms in a 1:1:1 ratio: KDS2010 120 mg, KDS2010 180 mg, and placebo. Randomization will consider stratification by region (Korea/USA). All subjects will undergo a 2-week run-in period prior to randomization to confirm eligibility based on adherence to lifestyle modification (documented reduction of ≥500 kcal/day and ≥150 minutes of physical activity per week for ≥50% of the run-in period).

The treatment period consists of 12 weeks of once-daily oral administration of the investigational product (IP), followed by a 1-week post-treatment safety follow-up (week 13). During treatment, subjects will visit the site at Weeks 4, 8, and 12, with a telephone visit at Week 2. Safety follow-up will be conducted by phone at Week 13.

The primary efficacy endpoint is the percentage change in body weight from baseline to Week 12. Secondary efficacy endpoints include the proportion of subjects achieving ≥5%, ≥10%, ≥15%, and ≥20% weight loss and changes in waist circumference, BMI, blood pressure (SBP/DBP), quality of life (IWQOL-Lite-CT), body composition (DEXA), lipid profile, glycemic parameters (HbA1c, fasting glucose, HOMA-IR), and liver steatosis. Exploratory endpoints assess the proportion of subjects with ≥25% weight loss, as well as changes in MAO-B specific activity and adiponectin levels.

Safety will be evaluated through monitoring of adverse events (AEs), laboratory tests, vital signs, ECGs, and psychological assessments, including the Columbia-Suicide Severity Rating Scale (C-SSRS) and Patient Health Questionnaire-9 (PHQ-9). Pharmacokinetic parameters (AUCtau, Cmax,ss, Cmin,ss, Cav,ss, Tmax,ss, t1/2, PTF, etc.) will be measured to assess systemic exposure to KDS2010.

Subjects must be adults (≥18 years), have a BMI ≥30 kg/m² or ≥27 kg/m² with at least one weight-related comorbidity, and demonstrate compliance with lifestyle modification during the run-in. Major exclusion criteria include recent significant weight change (≥5% within 12 weeks), use of anti-obesity drugs or MAO inhibitors, type 1 or 2 diabetes, bariatric surgery, uncontrolled hypertension, hepatic or renal dysfunction, significant psychiatric disorders, or suicidal ideation/attempts.

The total study duration is expected to be approximately 24 months from the IRB/IEC approval, with individual subject participation lasting up to 17 weeks. This trial aims to evaluate the safety, efficacy, and pharmacokinetic of KDS2010 for future development in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 years or older (or the legal age of adulthood in the respective country) as of the date of written consent
* Subjects with BMI ≥30 kg/m² or BMI ≥27 kg/m² with at least one weight-related comorbidity (hypertension, dyslipidemia, cardiovascular disease, obstructive sleep apnea) at screening and baseline

  * Hypertension: under treatment or have Systolic Blood Pressure (SBP) ≥130 mmHg or Diastolic Blood Pressure (DBP) ≥80 mmHg
  * Dyslipidemia: under treatment or LDL > 160 mg/dL or TG > 200 mg/dL or HDL < 40 mg/dL
  * Cardiovascular diseases (e.g., ischemic cardiovascular disease, NYHA Class I to III heart failure, Peripheral vascular disease (PVD), Abdominal aortic aneurysm (AAA), etc.)
  * Obstructive sleep apnoea
* Subjects who have documented a 500 kcal reduction/day in calorie intake and ≥150 minutes of physical activity/week for ≥50% of the time during the run-in period
* Subjects who have voluntarily provided written consent to participate after being informed about this clinical trial

Exclusion Criteria:

* Subjects with a weight change of 5% or more within 12 weeks before screening
* Subjects with less than 80% or more than 120% compliance during the Run-in period
* Subjects with obesity due to secondary causes (neurological disorders, endocrine disorders, genetic disorders, congenital disorders, etc.)
* Subjects with following medical history,

  * Type 1 or Type 2 diabetes
  * History of bariatric/metabolic surgery (e.g., adjustable gastric banding, intragastric balloon insertion, sleeve gastrectomy, Roux-en-Y gastric bypass, biliopancreatic diversion, duodenal switch) or planning to undergo such surgery during the study period
  * Heart failure classified as NYHA class IV
  * Subjects with a medical history of malignant tumors within 5 years prior to screening (however, subjects with successfully treated basal cell carcinoma, squamous cell carcinoma of the skin, thyroid cancer, or other carcinoma in situ, with no recurrence for more than 3 years, may be enrolled at the investigator's discretion)
  * Subjects with a medical history of hypersensitivity to MAO inhibitors
  * Subjects with a medical history of cerebrovascular disease (e.g., transient ischemic attack, stroke) within 12 weeks prior to baseline, or those hospitalized for unstable angina or congestive heart failure
  * Subjects with a history of depressive disorders or psychiatric disorders (e.g., schizophrenia, bipolar disorder, anxiety disorder) within 2 years prior to screening
* Subjects with a history of the following drug administration,

  -- Anti-obesity agents or weight-loss medications (including dietary supplements and herbal medicine) within 12 weeks before screening
  * Corticosteroids administered for 2 consecutive weeks or more within 12 weeks before screening (however, topical preparations, including inhalants, are allowed)
  * Treatment for hyperthyroidism or hypothyroidism at the time of screening (subjects on a stable dose and regimen for at least 12 weeks may be enrolled at the investigator's discretion)
  * MAO inhibitors within 2 weeks before baseline
  * Opioid medications (e.g., pethidine, Tramadol, Tapentadol) within 2 weeks before baseline
  * Serotonergic drugs within 2 weeks before baseline,

    * Selective Serotonin Reuptake Inhibitors (SSRI), ② Serotonin-Norepinephrine Reuptake Inhibitors (SNRI),

      * Tricyclic or Tetracyclic antidepressant, ④ Triazolopyridine antidepressant, ⑤ Selective serotonin (5-HT1) agonists (Sumatriptan, etc.), (However, amitriptyline ≤50 mg/day, trazodone ≤100 mg/day, citalopram ≤20 mg/day, sertraline ≤100 mg/day, paroxetine ≤30 mg/day are allowed; long half-life serotonergic drugs (e.g., fluoxetine) require at least a 5-week wash out period before enrollment),
  * Lithium, Bupropion, Lamotrigine, Ritonavir, Cyclobenzaprine, or St. John's wort within 2 weeks before baseline
  * Hypertension crisis-inducing drugs (e.g., oxymetazoline, phentermine, phenylephrine) within 2 weeks before baseline
  * Sympathomimetic agents (e.g., ephedrine, methylphenidate, amphetamine, methamphetamine, lisdexamfetamine) at the time of screening
  * Dextromethorphan at the time of screening
* Subjects who meet following criteria based on the tests conducted at Screening

  * Glycated hemoglobin (HbA1c) ≥6.5%
  * Hepatic impairment (Child-pugh class C)
  * AST or ALT > 2.5 X ULN
  * Total bilirubin >1.5 X ULN (however, >3.0 mg/dL is acceptable in cases of Gilbert syndrome)
  * Severe renal impairment (eGFR <30 mL/min/1.73 m² calculated using the MDRD formula*),

    * eGFR = 175 X (Serum creatinine)-1.154 X (Age)-0.203 X (0.742 (for females)) X (1.212 (for African Americans))
  * TSH >6.0 mIU/L or <0.4 mIU/L,
* Subjects with a lifetime history of suicide attempts
* Subjects with a PHQ-9 score of 10 or higher at screening
* Subjects who answer affirmatively to item 4 or 5 on the C-SSRS at screening
* Pregnant or breastfeeding women
* Females of childbearing potential and males who do not agree to use adequate contraception# until at least 2 weeks after the last dose of the IP or who plan to conceive during the study period,

  * Adequate contraception is defined as double contraception using both barrier methods (male condom or female condom) and one of the contraceptive methods ①-③.

    * Hormonal contraceptive (oral, injectable, implantable, etc.), ② Implantation of Intrauterine device (IUD) or intrauterine system (IUS), ③ Sterilization procedures or surgeries (bilateral tubal ligation, hysterectomy, vasectomy), ④ Complete abstinence: absolute abstinence is accepted if, in the investigator's judgment, the subject's age, occupation, lifestyle, or sexual orientation ensure compliance with contraception. However, periodic abstinence (calendar method, ovulation method, symptothermal method, etc.) withdrawal, and coitus interruptus are not considered adequate contraceptive methods.,
* Subjects who have participated in another clinical trial and received an investigational drug or device within 4 weeks prior to screening
* Other reasons (such as a medical history of alcohol or substance abuse) that the investigator deems the subject unsuitable for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Body Weight from Baseline | Baseline to Week 12
  The percentage change in body weight from baseline to Week 12 after administration of the investigational product (KDS2010).

SECONDARY OUTCOMES:
Proportion of Subjects with ≥5%, ≥10%, ≥15%, and ≥20% weight loss from baseline (%) | Baseline to Week 12
  Proportion (%) of subjects with ≥5%, ≥10%, ≥15%, and ≥20% weight loss at week 12 after IP administration compared to baseline
Change from baseline in Waist Circumference | Screening(Week -4 to -2), Run-in(Week -2), Baseline(Week 0), Week 4, 8, 12
  Waist circumference will be measured to the nearest 0.1 cm using a tape measure while the participant stands with feet approximately 25-30 cm apart, distributes body weight evenly, and exhales comfortably. Changes will be assessed up to Week 12.
Change from baseline in Body Mass Index (BMI) | Screening(Week -4 to -2), Run-in(Week -2), Baseline(Week 0), Week 4, 8, 12
  Change from baseline to Week 12 in BMI, calculated as weight in kilograms divided by height in meters squared (kg/m²).
Change from baseline in Systolic and Diastolic Blood Pressure | Screening(Week -4 to -2), Run-in(Week -2), Baseline(Week 0), Week 4, 8, 12, 13
  Change from baseline in systolic and diastolic blood pressure measured in mmHg.
Change from baseline in Impact of Weight on Quality of Life Questionnaire-Lite Clinical Trials version (IWQOL-Lite-CT) Total and Domain Scores | Baseline(Week 0), Week 12
  Change from baseline to Week 12 in the total score and domain-specific scores of the IWQOL-Lite-CT. IWQOL-Lite-CT is a questionnaire used to assess weight-related quality of life, consisting of 20 items. Each of the 20 items is evaluated on a scale of 0 to 5 points. Higher scores indicate better quality of life.
Change from baseline in Body Fat Composition via Dual-energy X-ray absorptiometry (DEXA) Scan | Baseline(Week 0), Week 12
  Change from baseline to Week 12 in percent body fat composition(changes in body fat mass and lean muscle mass) measured by DEXA scan.
Change from baseline in Lipid Profile | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12, 13
  Change from baseline in lipid parameters, including Total Cholesterol (TC), Triglycerides (TG), High-density lipoprotein cholesterol (HDL-C), Low-density lipoprotein cholesterol (LDL-C), Very low-density lipoprotein cholesterol (VLDL-C) and Free Fatty Acids.
Change from baseline in Glycemic Parameters: HbA1c (%) | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12, 13
  Change from baseline in Hemoglobin A1c (HbA1c) (percentage)
Change from baseline in Glycemic Parameters: Fasting Glucose (mg/dL) | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12, 13
  Change from baseline in fasting glucose levels (mg/dL).
Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline(Week 0), Week 12
  Change from baseline to Week 12 in HOMA-IR index. HOMA-IR is calculated using fasting insulin and fasting glucose levels to predict insulin resistance.
Change from baseline in Liver Steatosis (Abdominal CT) | Baseline(Week 0), Week 12
  Change from baseline to Week 12 in liver fat content assessed by Abdominal CT.

OTHER OUTCOMES:
Number of subjects with treatment-related Adverse Events (AEs) | Conducted from screening (Week -4 to -2) through Treatment (Week 0 to 12) and Follow-up (Week 13)
  AEs will be coded using MedDRA and assessed for severity and causality using CTCAE v5.0. The number of subjects affected and the incidence rates will be presented for each treatment group.
Change from baseline in laboratory test results | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12, 13
  Laboratory parameters including routine hematology, blood chemistry, urinalysis, lipid, coagulation, hormone will be measured. Change from baseline will be analyzed.
Change from baseline in pulse rate | Screening(Week -4 to -2), Run-in(Week -2), Baseline(Week 0), Week 4, 8, 12, 13
  Pulse rate will be measured in beats per minute.
Change from baseline in body temperature | Screening(Week -4 to -2), Run-in(Week -2), Baseline(Week 0), Week 4, 8, 12, 13
  Body temperature will be measured using a standard thermometer.
Change from baseline in Electrocardiogram(ECG) | Screening(Week -4 to -2), Week 12, 13
  For ECG results, the proportion of subjects whose status changed from 'Normal or Abnormal Not Clinically Significant (Abnormal NCS)' before the IP administration to 'Abnormal Clinically Significant (Abnormal CS)' after IP administration will be summarized and presented in a table.
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) total score | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12
  C-SSRS is used to assess the risk of suicide through interviews with the subject. The scores of each question are summed to range from 0 to 25 points. If "yes" from questions 4 or 5, categorize a subject as high-risk, requiring further evaluation, while other scores indicate a lower risk.
Change from baseline in Patient Health Questionnaire-9 (PHQ-9) | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12
  The PHQ-9 is a validated self-report tool used to screen for and assess the severity of depressive symptoms. It consists of nine items, each rated on a 4-point scale from 0 ("not at all") to 3 ("nearly every day"), with a total possible score ranging from 0 to 27. Higher scores indicate greater severity of depressive symptoms.
Proportion of Subjects with ≥25% Weight Loss at Week 12 | Baseline to Week 12
  Proportion (%) of subjects with ≥25% weight loss at week 12 after IP administration compared to baseline.
Percentage Change in Monoamine Oxidase B (MAO-B) Specific Activity | Baseline(Week 0), Week 12
  Percentage change in MAO-B specific activity compared to baseline (%)
Percentage Change in Adiponectin Levels | Screening(Week -4 to -2), Baseline(Week 0), Week 4, 8, 12, 13
  Percentage change in Adiponectin compared to baseline (%)
Pharmacokinetic Parameters: Area Under the Plasma Concentration-Time Curve over the dosing interval (τ) (AUCtau) at steady-state | Baseline(Week 0), Week 4, 8, 12
  AUCtau is the area under the plasma concentration-time curve over the dosing interval (τ) at steady-state, and it reflects the extent of drug exposure within a dosing cycle.
Pharmacokinetic Parameters: Peak Plasma Concentration at Steady State (Cmax,ss) | Baseline(Week 0), Week 4, 8, 12
  The highest plasma drug concentration observed during a dosing interval at steady-stat
Pharmacokinetic Parameters: Minimum Plasma Concentration at Steady State (Cmin,ss) | Baseline(Week 0), Week 4, 8, 12
  The lowest plasma drug concentration during a dosing interval at steady-state, usually occurring right before the next dose.
Pharmacokinetic Parameters: Average Plasma Concentration at Steady State (Cav,ss) | Baseline(Week 0), Week 4, 8, 12
  The average plasma concentration over the dosing interval at steady-state. Calculated as: Cav, ss = AUCtau/τ
Pharmacokinetic Parameters: Time to Maximum Plasma Concentration at Steady State (Tmax,ss) | Baseline(Week 0), Week 4, 8, 12
  The time taken to reach the maximum plasma concentration after dosing at steady-state.
Pharmacokinetic Parameters: Terminal Elimination Half-life (t1/2) | Baseline(Week 0), Week 4, 8, 12
  The time required for the plasma concentration of the drug to decrease by half.
Pharmacokinetic Parameters: Peak-Trough Fluctuation at Steady State (PTF) | Baseline(Week 0), Week 4, 8, 12
  A measure of the fluctuation between the peak (Cmax,ss) and trough (Cmin,ss) plasma concentrations during a dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sangwook Kim, Chief Executive Officer, Study Director — NeuroBiogen Co., Ltd
Locations (3):
- South Korea (3):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kangbuk Samsung Medical Center, Seoul, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No